CLINICAL TRIAL: NCT00525915
Title: An Oxaliplatin-Based Phase II Randomized Study of Induction Chemotherapy Followed by Preoperative Chemoradiotherapy or Preoperative Chemoradiotherapy in Patients With Resectable Esophageal or Gastroesophageal Carcinoma
Brief Title: Oxaliplatin-Based Chemotherapy and Chemoradiotherapy or Chemoradiotherapy in Esophageal or Gastroesophageal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0703
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Esophageal Cancer; Gastroesophageal Cancer
Keywords: Esophageal Cancer; Gastroesophageal Cancer; Gastroesophageal Junction; Radiation Therapy; 5-Fluorouracil; 5-FU; Adrucil; Efudex; Oxaliplatin
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Fluorouracil; Oxaliplatin; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Chemo with Radiation Treatment (Experimental): For 5 weeks, Chemo of 5-FU 250 mg/m^2 intravenous (IV) over 24 hours for 5 days weekly with Oxaliplatin 40 mg/m^2 IV daily over 2 hours, and Radiation treatment every weekday; then surgery.
  Interventions: Drug: 5-Fluorouracil; Drug: Oxaliplatin; Radiation: Radiation Therapy; Procedure: Surgery
- Arm B: Pre-Op Chemo + Chemo with Radiation Treatment (Experimental): Pre-Operative Chemo 5-FU 2.2 mg/m^2 IV continuous infusion over 48 hours start on day 1 and 15, and Oxaliplatin 100 mg/m^2 IV on day 1 and 15; followed by Surgery + Chemo with Radiation Therapy (same as Arm A)
  Interventions: Drug: 5-Fluorouracil; Drug: Oxaliplatin; Radiation: Radiation Therapy; Procedure: Surgery

INTERVENTIONS:
Drug: 5-Fluorouracil — Arm A = 250 mg/m^2 IV over 24 hours for 5 days weekly for 5 weeks.
  Arm B = 2.2 mg/m^2 IV over 48 hours on days 1 and 15.
  Other Names: 5-FU; Adrucil; Efudex
Drug: Oxaliplatin — Arm A: 40 mg/m^2 IV daily over 2 hours for 5 weeks
  Arm B: 100 mg/m^2 IV on Day 1 and 15
  Other Names: Eloxatin
Radiation: Radiation Therapy — Radiation treatment every weekday for 5 weeks.
  Other Names: RT; XRT
Procedure: Surgery — Surgical removal of the primary tumor and lymph nodes following completion of disease status evaluation post chemotherapy and radiation treatments.

SUMMARY:
The goal of this clinical research study is to learn if a combination of the investigational drug oxaliplatin with 5-Fluorouracil (5-FU) (given at the same time as radiation therapy) is as effective as a combination of these two drugs given before and during radiation therapy in the treatment of esophageal or gastroesophageal cancers. The safety of these combinations of therapy will also be compared.

Objectives:

Primary objective:

Compare the Pathologic Complete Response rate and % of patients with <50% residual cancer in the resected surgical specimen between Arms A and B.

Secondary objectives:

1. Compare 1-year and 3-year survival rates, median survival time, R0 resection rates, safety, and local plus systemic relapse rates between Arms A and B
2. Perform exploratory correlative studies on blood, adjacent normal and cancer tissue to assess predictive markers of response and outcome.
3. Evaluate the joint effects, including possible interactive effects, of proton-versus-photon therapy and treatment arm on overall survival, R0 resection rates, safety, and local plus systemic relapse rates.

DETAILED DESCRIPTION:
Oxaliplatin and 5-FU are chemotherapy drugs that are commonly used to treat certain kinds of cancers. 5-FU is designed to prevent cells from making DNA that is necessary for cell growth. This disrupts the growth of the cancer cells, which causes the cancer cells to start to die. Oxaliplatin is designed to damage DNA that is already formed.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of two groups. Participants in the first group (Arm A) will receive chemotherapy with radiation treatment. Participants in the second group (Arm B) will receive chemotherapy first then chemotherapy with radiation treatment. The chemotherapy that will be used in this study includes 5-FU and oxaliplatin. Arm B is 8 weeks longer than Arm A. Your doctor will discuss with you whether you will receive proton or photon radiation. If you receive proton radiation, it will be given in a building that is about a 5 minute drive from the main MD Anderson radiation clinic.

All participants will have had a routine upper gastrointestinal tract endoscopy and biopsy with endoscopic ultrasound examination before receiving treatment on this study. However, once you start on this study, the upper gastrointestinal tract endoscopy will be repeated before the 2nd cycle of induction chemotherapy Arm B (if needed), before chemoradiation, and before surgery. This procedure involves examination of the esophagus, stomach, and duodenum by a flexible tube. Biopsies will be taken as necessary.

Arm A:

If you are assigned to Arm A, you will receive treatment with 5-FU over 24 hours for 5 days each week for 5 weeks. It will be given as an infusion into a vein using a portable pump. This will start on Day 1 (Monday) and will continue until Day 5 (Friday) of each radiotherapy week for 5 weeks. You will need to carry this pump with you for about 96 hours. The pump is about the size of a personal compact disc player. You will also receive oxaliplatin as an infusion into a vein over 2 hours on Day 1. This will be repeated on Days 8, 15, 22, and 29. During this time you will receive radiation therapy every weekday for 5 weeks.

If the cancer gets worse or you experience intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

Each week while you are receiving chemoradiotherapy, around 1 tablespoon of blood will be drawn for routine tests. Between 5-6 weeks after the completion of chemoradiotherapy, the stage of the cancer will be evaluated. This includes drawing blood (about 1 tablespoon) for routine tests, an Electrocardiography (ECG), a Physical Fitness Testing (PFT), a computed tomography (CT) of the abdomen and chest (when necessary), a Positron emission tomography (PET) or PET/CT scan, and an upper GI endoscopy with biopsies and checking the status of your abdominal disease (if necessary).

When the evaluation of the status of your disease is complete, surgical removal of the primary tumor and lymph nodes will be attempted. All participants with no spreading disease, who are physically able to have surgery and have disease that is judged to be removable will be eligible for surgery. The tube (J-tube) will be left in your body for at least 8 weeks after the surgery to supplement your nutrition.

Arm B:

If you are assigned to Arm B, you will receive a starting (induction) course of chemotherapy before radiation therapy ever starts. You will receive 5-FU over 48 hours as an infusion into a vein using a portable pump. This will start on Day 1 and will continue over 48 hours. This will be repeated on Day 15 for another 48 hours. You will need to carry this pump with you at all times from Days 1-2 and Days 15-16. The pump is about the size of a personal compact disc player. You will also receive oxaliplatin as an infusion into a vein over 2 hours on Days 1 and 15.

One cycle is equal to 28 days, which includes 2 doses of 5-FU and oxaliplatin given on Day 1 and Day 15. Treatment is always followed by 12 days of recovery. You will receive a maximum of 2 cycles (4 doses of 5-FU and oxaliplatin).

After the first and second cycles, you will be given a full physical exam, upper GI x-rays if necessary, about 1 tablespoon of blood will be drawn for routine blood tests, and if needed, a CT scan of the abdomen and chest will be performed. You will have a PET scan or PET CT scan and upper GI endoscopy with biopsy (if needed) before the start of Cycle 2 and after the end of Cycle 2. If the disease has not gotten worse after the 1st cycle of induction chemotherapy, you will receive the 2nd cycle. An upper gastrointestinal tract endoscopy and biopsy will be performed. If the disease gets worse at any stage, you will go straight to chemoradiotherapy. If the disease starts to spread, you will be taken off study and your doctor will discuss other treatment options with you.

You will begin to receive chemoradiotherapy no more than 12 days after you complete the last dose of induction chemotherapy. You will receive treatment with 5-FU over 24 hours for 5 days each week for 5 weeks. It will be given as an infusion into a vein using a portable pump. This will start on Day 1 (Monday) and will continue until Day 5 (Friday) of each radiotherapy week for 5 weeks. You will need to carry this pump with you at all times for about 96 hours. You will also receive oxaliplatin as an infusion into a vein over 2 hours on Day 1. This will be repeated on Days 8, 15, 22, and 29. During this time you will receive radiation therapy every weekday for 5 weeks.

If the cancer gets worse or you experience intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

Each week while you are receiving chemoradiotherapy, around 1 tablespoon of blood will be drawn for routine tests. Between 5-6 weeks after the completion of chemoradiotherapy, the stage of the cancer will be evaluated. This includes drawing blood (about 1 tablespoon) for routine tests, an ECG, a PFT, a CT of the abdomen and chest (when necessary), a PET Scan or PET CT Scan, and an upper GI endoscopy with biopsies and checking the status of your abdominal disease (if necessary).

When the evaluation of the status of your disease is complete, surgical removal of the primary tumor and lymph nodes will be attempted. All participants with no spreading disease, who are physically able to have surgery and have disease that is judged to be removable will be eligible for surgery. The a tube (J-tube) will be left in your body for at least 8 weeks after the surgery to supplement your nutrition.

Arms A and B:

You will be asked to fill out side effect sheets throughout your participation in this research study. You will be asked questions regarding nausea, hair loss, fatigue, meals, and other questions regarding your daily activities. You will be asked to keep a daily calendar while receiving therapy of any type.

You will be asked to come for follow-up visits at MD Anderson at 3, 6, 9, and 12 months after surgery and then every 6 months for 2 years, and then once a year for 2 years. At these visits, you will have a full physical exam, and about 1 tablespoon of blood drawn for routine tests and a CEA test (carcinoembryonic antigen - a protein made by cancer and normal cells) if your CEA level was high in the past. You will also have a PET scan, PET CT scan, or CT of the chest and abdomen. You will have an upper GI endoscopy with biopsies 3 months after surgery and at other follow-up visits if needed. You may have a CT of the chest and abdomen at the 3 month visit if needed.

This is an investigational study. Oxaliplatin is an investigational drug and is not approved in the US for use in the treatment of esophageal and gastroesophageal cancer. The combination of these 2 drugs (oxaliplatin + 5-FU) is investigational. All procedures are standard of care. A total of up to 126 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Local regional carcinoma of the thoracic esophagus (squamous cell or adeno) or gastroesophageal junction.
2. Patients with T1N1, and T2-3 with any N (M1a only) will be eligible.
3. Normal liver (serum glutamic-pyruvic transaminase (SGPT) < 56µL, Total Bilirubin <1.5 mg/dL), kidney (Creatinine <1.75 mg/dL), and bone marrow functions (AGN >1,500µL, platelet count >100,000/µL).
4. Performance status 0 or 1.
5. Signed informed consent by the investigator or their designee and patient.
6. Medically fit for surgery.
7. No Celiac (except for the GE junction cancers), supraclavicular, or paraaortic nodal enlargement unless biopsy negative.
8. None of the celiac nodes should be larger than 2 cm
9. Male or Female but both sexes must practice adequate contraception while on therapy
10. >/=18 years but less than 76 years
11. No known allergy to any of the study drugs.
12. No prior therapy for this cancer.
13. No significant cancer (defined as non-melanomatous skin cancers and treated cervical cancers) within the past 5 years
14. New York Heart Association (NYHA) I and II

Exclusion Criteria:

1. Patients with T1N0, T4, or M1b cancer will be excluded
2. Significant comorbid conditions (defined as uncontrolled diabetes, active angina or heart failure, uncontrolled hypertension, or active psychiatric condition that prevents consistent participation and compliance).
3. More than grade 1 neuropathy
4. Unable to comprehend the requirements of the study or comply with it.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Ajani, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Shimodaira Y, Slack RS, Harada K, Chen HC, Sagebiel T, Bhutani MS, Lee JH, Weston B, Elimova E, Lin Q, Amlashi FG, Mizrak Kaya D, Blum MA, Roth JA, Swisher SG, Skinner HD, Hofstetter WL, Rogers JE, Mares J, Thomas I, Maru DM, Komaki R, Walsh G, Ajani JA. Influence of induction chemotherapy in trimodality therapy-eligible oesophageal cancer patients: secondary analysis of a randomised trial. Br J Cancer. 2018 Feb 6;118(3):331-337. doi: 10.1038/bjc.2017.423. Epub 2017 Dec 12. PMID 29235564
- [Derived] Harada K, Wang X, Shimodaira Y, Sagebiel T, Bhutani MS, Lee JH, Weston B, Elimova E, Lin Q, Amlashi FG, Mizrak Kaya D, Lopez A, Blum Murphy MA, Roth JA, Swisher SG, Skinner HD, Hofstetter WL, Rogers JE, Thomas I, Maru DM, Komaki R, Walsh G, Ajani JA. Early Metabolic Change after Induction Chemotherapy Predicts Histologic Response and Prognosis in Patients with Esophageal Cancer: Secondary Analysis of a Randomized Trial. Target Oncol. 2018 Feb;13(1):99-106. doi: 10.1007/s11523-017-0540-3. PMID 29218623
- [Derived] Ajani JA, Xiao L, Roth JA, Hofstetter WL, Walsh G, Komaki R, Liao Z, Rice DC, Vaporciyan AA, Maru DM, Lee JH, Bhutani MS, Eid A, Yao JC, Phan AP, Halpin A, Suzuki A, Taketa T, Thall PF, Swisher SG. A phase II randomized trial of induction chemotherapy versus no induction chemotherapy followed by preoperative chemoradiation in patients with esophageal cancer. Ann Oncol. 2013 Nov;24(11):2844-9. doi: 10.1093/annonc/mdt339. Epub 2013 Aug 23. PMID 23975663
- See also: UT MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 01, 2005 to June 20, 2011. All recruitment done at UT MD Anderson Cancer Center.
Groups:
- Arm A: Chemo With Radiation Treatment: For 5 weeks, Chemotherapy (Chemo) of 5-Fluorouracil (5-FU) 250 mg/m^2 intravenous (IV) over 24 hours for 5 days weekly with Oxaliplatin 40 mg/m^2 IV daily over 2 hours, and Radiation treatment every weekday; then surgery.
- Arm B: Pre-Op Chemo + Chemo With Radiation Treatment: Pre-Operative Chemo 5-FU 2.2 mg/m^2 IV continuous infusion over 48 hours start on day 1 and 15, and Oxaliplatin 100 mg/m^2 IV over 2 hours on day 1 and 15; followed by Surgery + Chemo with Radiation Therapy (same as Arm A)
Period: Overall Study
Arm/Group | Arm A: Chemo With Radiation Treatment | Arm B: Pre-Op Chemo + Chemo With Radiation Treatment
Started | 63 | 63
Completed | 55 (Participants who underwent surgery.) | 54
Not Completed | 8 | 9
Not completed — Non-Compliance | 0 | 1
Not completed — Disease Progression | 5 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Refused Surgery | 1 | 2
Not completed — Unrelated illness | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of the 126 randomized, 2 participants in Arm A declined therapy after randomization; and 13 (6 in Arm A and 7 in Arm B) experienced treatment failure before surgery leaving 55 in Arm A participants and 54 in Arm B who underwent surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Chemo With Radiation Treatment | Arm B: Pre-Op Chemo + Chemo With Radiation Treatment | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 74] | 60 [27 to 75] | 60 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 59 | 59 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 61 | 63 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 60 | 60 | 120
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 63 | 126

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: Pathologic Complete Response rate: percentage of participants with response reported as Pathologic complete response (pathCR) following surgery. Once surgery performed, response to therapy judged in surgical specimen with three possible categories reported: 1) Pathologic complete response (no residual cancer in the specimen); 2) <50% of residual cells in the surgical specimen; or 3) >50% of cells in the surgical specimen. Upon recovery from chemoradiation (Chemo), surgery follows approximately 5-6 weeks later with response assessment. Arm A schedule consists of 6 weeks of Chemo +XRT, followed by 5-6 weeks of rest, followed by surgery. Arm B schedule consist of 8 weeks of Chemo, followed by 6 weeks of Chemo +XRT, followed by 5-6 weeks of rest, followed by surgery. In particular, Arm B is 8 weeks longer than Arm A.
Time Frame: Surgery post chemotherapy (approximately 10-11 weeks)
Population: Participants who had surgery were reported for the pathCR rate assessment in this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Chemo With Radiation Treatment | Arm B: Pre-Op Chemo + Chemo With Radiation Treatment
Number analyzed (Participants) | 55 | 54
percentage of participants | 13 | 26

ADVERSE EVENTS:
Time Frame: Adverse events recorded for all participants from randomization until 30 days following last dose of study treatment (including withdrawal because of toxicity). Overall active study period was from April 2005 to July 2012.
Arm/Group | Arm A: Chemo With Radiation Treatment | Arm B: Pre-Op Chemo + Chemo With Radiation Treatment
Serious Adverse Events (participants affected / at risk) | 10/63 | 7/63
Other Adverse Events (participants affected / at risk) | 63/63 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Chemo With Radiation Treatment (N=63) | Arm B: Pre-Op Chemo + Chemo With Radiation Treatment (N=63)
DEHYDRATION (Gastrointestinal disorders) | 2 (2) | 1 (1)
NAUSEA/VOMITING (Gastrointestinal disorders) | 3 (3) | 0 (0)
FEVER (Investigations) | 2 (2) | 1 (1)
Gastrointestinal (GI) BLEED (Gastrointestinal disorders) | 1 (1) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 2 (2)
DYSPHAGIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Chemo With Radiation Treatment (N=63) | Arm B: Pre-Op Chemo + Chemo With Radiation Treatment (N=63)
ANOREXIA (Gastrointestinal disorders) | 46 (46) | 43 (43)
DERMATITIS (RADIATION) (Skin and subcutaneous tissue disorders) | 23 (23) | 16 (16)
FATIGUE (General disorders) | 54 (54) | 51 (51)
LEUKOPENIA (Blood and lymphatic system disorders) | 23 (23) | 32 (32)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
ANEMIA (Blood and lymphatic system disorders) | 51 (51) | 50 (50)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 15 (15) | 31 (31)
VOMITING (Gastrointestinal disorders) | 28 (28) | 16 (16)
DYSPHAGIA (Respiratory, thoracic and mediastinal disorders) | 48 (48) | 42 (42)
NEUROPATHY SENSORY (Nervous system disorders) | 37 (37) | 27 (27)
MYALGIA (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (10)
DIARRHEA (Gastrointestinal disorders) | 29 (29) | 15 (15)
ODYNOPHAGIA (Respiratory, thoracic and mediastinal disorders) | 24 (24) | 17 (17)
DEHYDRATION (General disorders) | 5 (5) | 2 (2)
INCREASE Alanine Aminotransferase (ALT) (Hepatobiliary disorders) | 23 (23) | 19 (19)
INCREASE Aspartate Aminotransferase (AST) (Hepatobiliary disorders) | 21 (21) | 28 (28)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
FEVER (Investigations) | 12 (12) | 6 (6)
CHILLS (General disorders) | 3 (3) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 36 (36) | 24 (24)
Gastroesophageal reflux disease (GERD) (Gastrointestinal disorders) | 38 (38) | 30 (30)
MUCOSITIS (Gastrointestinal disorders) | 15 (15) | 8 (8)
RED, WATERY and BURNING EYES (Eye disorders) | 9 (9) | 4 (4)
ALOPECIA (Immune system disorders) | 2 (2) | 6 (6)
DIZZINESS (Nervous system disorders) | 23 (23) | 15 (15)
INSOMNIA (Nervous system disorders) | 41 (41) | 33 (33)
ABDOMINAL PAIN (General disorders) | 5 (5) | 4 (4)
PAIN (General disorders) | 12 (12) | 13 (13)
BACK PAIN (General disorders) | 9 (9) | 10 (10)
HEADACHE (Nervous system disorders) | 11 (11) | 6 (6)
SUBSTERNAL CHEST PAIN (General disorders) | 6 (6) | 2 (2)
CHEST PAIN (General disorders) | 4 (4) | 3 (3)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 11 (11)
HICCUPS (General disorders) | 20 (20) | 24 (24)
COUGH (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 14 (14)
TINNITUS (Ear and labyrinth disorders) | 8 (8) | 5 (5)
TASTE CHANGE (General disorders) | 25 (25) | 26 (26)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
ESOPHAGITIS (Gastrointestinal disorders) | 19 (19) | 14 (14)
DERMATITIS (Skin and subcutaneous tissue disorders) | 26 (26) | 37 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No